CLINICAL TRIAL: NCT00659672
Title: Effect of Whey Protein on Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: David J. Baer, Ph.D, Principal Investigator, USDA-ARS
Organization: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 2007-384
Record Dates: First submitted 2008-04-14; First posted 2008-04-16 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2011-02

CONDITIONS: High Blood Pressure
Keywords: hypertension; prehypertension; high blood pressure; blood pressure; heart disease
MeSH Terms: conditions — Hypertension; Prehypertension; Heart Diseases | interventions — Whey Proteins; Soybean Proteins; Carbohydrates

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Whey Protein — 40 grams per day Whey Protein
Dietary Supplement: Soy Protein — 40 grams per day soy protein
Dietary Supplement: Control (carbohydrate) — 40 grams per day maltodextrin

SUMMARY:
The purpose of this study is to determine if consumption of whey protein, compared with soy protein or a carbohydrate food decreases blood pressure along with reducing risk factors for heart disease.

DETAILED DESCRIPTION:
Several lines of evidence suggest that consumption of dairy foods, and specifically whey protein, may reduce blood pressure. This proposed study is designed investigate the effect of whey protein compared to another protein source.

Since blood pressure is a recognized risk factor for cardiovascular disease, if there is clear evidence that whey protein reduces blood pressure, dietary recommendations may be made regarding whey protein intake. However, dietary recommendations to consume whey protein as a means to improve health status must be science-based. Results from this study will provide a scientific basis for dietary recommendations regarding whey protein intake.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 42 kg/m2
* Fasting glucose < 126 mg/dl
* Blood pressure > 120/80 and < 160/100 mm Hg [based two measurements collected on separate days]

Exclusion Criteria:

* Use of prescription or over-the-counter medications that alter blood pressure.
* Presence of kidney disease, liver disease, gout, certain cancers, thyroid disease, gastrointestinal, other metabolic diseases, or malabsorption syndromes.
* Women who have given birth during the previous 12 months.
* Pregnant women or women who plan to become pregnant or become pregnant during the study.
* Lactating women.
* Type 2 diabetes requiring the use of oral antidiabetic agents or insulin.
* History of eating disorders or other dietary patterns which are not consistent with the dietary intervention (e.g., vegetarians, very low fat diets, high protein diets).
* Volunteers who routinely participate in "heavy" exercise or volunteers who initiate an exercise program during the study.
* Volunteers who have lost 10% of body weight within the last 12 months.
* Use of vitamin and mineral supplements or antacids containing magnesium or calcium.
* Use of prescription or over-the-counter antiobesity medications or supplements (e.g., phenylpropanalamine, ephedrine, caffeine, during and for at least 6 months prior to the start of the study) or history of a surgical intervention for obesity.
* Active cardiovascular disease (such as heart attack or procedure within the past three months or participation in a cardiac rehabilitation program within last three months, stroke or history/treatment for transient ischemic attacks in the past three months, or documented history of pulmonary embolus in past six months).
* Smokers or other tobacco users (during the 6 months prior to the start of the study).
* Known (self-reported) allergy or adverse reaction to dairy products (including lactose) or soy.
* Unable or unwilling to give informed consent or communicate with study staff.
* Self-report of alcohol or substance abuse within the past twelve months and/or current acute treatment or rehabilitation program for these problems (Long-term participation in Alcoholics Anonymous is not an exclusion.)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol.

Ages: 28 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
systolic and diastolic blood pressure | monthly

SECONDARY OUTCOMES:
Hormones,lipoproteins, and inflammation | monthly

CONTACTS AND LOCATIONS:
Overall Officials: David J Baer, Ph.D., Principal Investigator — USDA-ARS, Beltsville Human Nutrition Research Center
Locations (1):
- USDA Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States